CLINICAL TRIAL: NCT00163176
Title: Value of FLT-PET Before and During Radiotherapy in Head and Neck Tumors
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 049
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Head and Neck Neoplasms
Keywords: cell proliferation; PET; radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Tumor cell proliferation and repopulation contribute to resistance to radiotherapy in head and neck cancer. Up to now, this characteristic is mostly assessed using biopsies acquired during inspection under general anaesthesia before treatment.

18F-FLT-PET (positron emission tomography) is a non-invasive imaging method showing areas of active proliferation. The aim of this study is to assess the value of the functional information gained by 18F-FLT-PET for radiotherapy planning and early tumor response assessment.

Prior to radiotherapy, a planning CT-scan and a 18F-FLT-PET scan are acquired. After approximately two weeks of radiotherapy a further PET scan is obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Stage II - IV squamous cell carcinoma of the head-and-neck region, treated with radiotherapy or radiochemotherapy with curative intent.
2. 18 years or older
3. Informed consent

Exclusion Criteria:

1. Patients who have undergone surgery as primary tumor therapy.
2. Patients treated with palliative intent.
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage II-IV squamous cell carcinoma of the head and neck
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Correlation of 18F-FLT-PET-signal changes before and during therapy with treatment outcome (clinical response and local tumor control) | 1 year

SECONDARY OUTCOMES:
Evaluation of the value of the functional information gained by 18F-FLT-PET regarding the definition of the planning target volume (PTV) for radiotherapy. | 2 months
Measurement of 18F-FLT-PET-signal changes during radiotherapy or radiochemotherapy. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Johannes HA Kaanders, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen, Department of Radiotherapy, Nijmegen, Gelderland, Netherlands